CLINICAL TRIAL: NCT00322296
Title: A Phase II Trial to Evaluate the Efficacy of Topical Bexarotene Gel in Patients With Parapsoriasis: a Topical Chemoprevention Strategy for Cutaneous T-cell Lymphoma.
Brief Title: Phase II Trial to Evaluate the Efficacy of Topical Bexarotene Gel in Patients With Parapsoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The response rate (5/8) had reached a statistical significant endpoint.
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Ligand Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-031
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2006-05

CONDITIONS: Parapsoriasis
Keywords: Parapsoriasis; Cutaneous T-cell lymphoma; Mycosis fungoides; Bexarotene; Retinoids
MeSH Terms: conditions — Parapsoriasis; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Bexarotene; Gels

INTERVENTIONS:
Drug: Bexarotene 1% gel

SUMMARY:
Parapsoriasis is a term that refers to a precursor stage of cutaneous T-cell lymphoma (CTCL)/mycosis fungoides(MF). Complete responses (clearing) of early presentations of CTCL/MF have been shown to be associated with long-term survival and cure. Induction of a complete response in parapsoriasis, therefore, would seem to be a desirable therapeutic endpoint. Bexarotene 1% gel has been approved for treatment of cutaneous T-cell lymphoma (mycosis fungoides). The goal of this study is to evaluate the tolerability, safety and efficacy of bexarotene 1% gel in patients with parapsoriasis.

DETAILED DESCRIPTION:
Parapsoriasis is a term that refers to a red, scaling (papulosquamous) eruption on the skin characterized by its distribution (trunk and proximal extremities), asymptomatic nature and chronic course. Histologically, parapsoriasis is characterized by variable degrees of parakeratosis and epidermal spongiosis with a superficial, sparse, patchy, lichenoid infiltrate of lymphocytes and varying degrees of epidermal involvement (epidermotropism). No definitive studies have defined its etiology or epidemiology.

Historically, the term "parapsoriasis" was introduced into the dermatology literature by Brocq in 1902. Brocq used the term to clinically characterize a variety of papulosquamous eruptions that were first reported in the late 19th century. In 1905, he attempted to categorize parapsoriasis in relationship to other papulosquamous diseases of the skin. In his model, Brocq delineated a relationship between some variants of parapsoriasis (parapsoriasis en plaques or large plaque parapsoriasis) and mycosis fungoides or cutaneous T-cell lymphoma (CTCL). The first cases of mycosis fungoides (MF) were reported early in the 19th century. Progressive stages of MF ("premycotic" patch phase, plaque phase and tumor phase) were defined later in the 19th century, while the neoplastic nature of the disease remained unknown. Brocq's model sought to emphasize clinical similarities between some variants of parapsoriasis (large plaque) and early, patch phase MF.

Immunohistochemical (IHC) studies have demonstrated that parapsoriasis shares a similar immunophenotype with early stage CTCL in that the lymphocytic infiltrate is predominantly composed of CD4 lymphocytes. Polymerase chain reaction (PCR)- based T-cell receptor (TCR) gene rearrangement studies have demonstrated that parapsoriasis is a lymphoproliferative disorder characterized by the detection of clonal populations of T-cells, as is CTCL. Knowledge of the natural history of parapsoriasis stems from a series of longitudinal outcome studies published over the last 40 years. Progression to unequivocal CTCL ranged from 0% to 35% of parapsoriasis cases. Typically, cases associated with progression to CTCL tend to have larger plaques with clinical features of atrophy and/or poikiloderma.

Based on the clinicopathologic similarities of parapsoriasis and early stage CTCL, the exact nosology of parapsoriasis has been challenged, with a hypothesis that all variants of parapsoriasis (large plaque, small plaque and digitate) are synonymous with early MF. Nevertheless, parapsoriasis is recognized as a distinct precursor stage (T0N0M0) in the TNM staging schema of CTCL. T0 CTCL is defined by the presence of lesions clinically and/or histologically suggestive of CTCL.

No definitive studies have been published regarding therapy of parapsoriasis. When treated, most patients are initiated empirically on topical steroids or phototherapy. Typically, patients will have partial responses and/or relapse off any therapy. A rational therapeutic strategy for parapsoriasis is lacking because there are no longitudinal studies that correlate treatment response and impact on progression to CTCL.

Bexarotene is a resinoid, a subclass of retinoids that binds preferentially to nuclear retinoic X receptors (RXR), and has therapeutic activity in CTCL. Bexarotene 1% gel has been approved for treatment of CTCL and found to have up to a 63% response rate in Stage Ia to IIa CTCL. The goal of this study was to evaluate the tolerability, safety and efficacy of bexarotene 1% gel in patients with parapsoriasis and to evaluate the anti-tumor host response in pre- and post-treatment skin biopsies.

ELIGIBILITY:
Inclusion Criteria:

* A clinical and histologic diagnosis of parapsoriasis (T0 CTCL)
* Age 18 years or older.
* Acceptable laboratory studies
* Must be free of serious concurrent illness.
* Women of child-bearing potential must have negative serum pregnancy test prior to the initiation of treatment.

Exclusion Criteria:

* Topical or systemic therapies within four weeks of entry in the study.
* Participation in any other investigational drug study within thirty days of entry in this study.
* Oral retinoid therapy for any indication within three months of entry in the study.
* Participation in any other study using topical retinoid therapy.
* Pregnancy or active breast-feeding.
* Serious known concurrent medical illness or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2001-04; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoints (outcome) are the skin lesion responses determined by the Composite Assessment of Index Lesion Disease Severity following up to sixteen weeks of treatment

SECONDARY OUTCOMES:
Secondary efficacy endpoints (outcomes) include the disease response to treatment as determined by percentage of total body surface area involvement and physician global assessment following up to sixteen weeks of treatment.
Also, antitumor host response as determined by immunohistochemistry in pre and post treatment skin biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart R. Lessin, M.D., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States